CLINICAL TRIAL: NCT05391386
Title: Evaluation of Failure Rate of Molar Tube With a Modified Bonding Technique: A Randomized Clinical Trial
Brief Title: Evaluation of Failure Rate of Molar Tube With a Modified Bonding Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Nawar Mohammed Hasan, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 601422
Record Dates: First submitted 2022-05-21; First posted 2022-05-26 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Molar Tube Bonding
Keywords: molar tube; failure rate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (No Intervention)
- modified (Experimental)
  Interventions: Procedure: modified bonding technique

INTERVENTIONS:
Procedure: modified bonding technique — adding a layer of compomer adhesive at the molar/tube interface.
  Arms: modified

SUMMARY:
Comparing between the failure rates of molar tubes bonded with conventional bonding technique using resin adhesive and the alternative bonding technique using compomer (containing glass ionomer) adhesive by adding a layer of compomer adhesive at the molar/tube interface.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring fixed appliance orthodontic treatment (with no previous orthodontic treatment).
2. Patients aged >12 years with full permanent dentition (excluding third molars).
3. Intact buccal enamel surface of the molars without any of the following:

   * Caries, abrasion, or any other crown defect (like hypoplasia).
   * Pretreatment chemical agents.
   * Restorations or fractures.
   * Morphological modifications or other crown alterations.
4. Patients who have the desire and ability to comply with the trial protocol.

Exclusion Criteria:

1. Treatments with planned extraction of first permanent molars.
2. Occlusal interference that prevents correct position of molar tube.
3. Patients with a craniofacial anomaly (like cleft lip and palate) and/or require orthognathic surgery.
4. Patients that require extra-oral or intra-oral anchorage device (headgear, palatal arch, lingual arch) or expander (quad-helix, hyrax).
5. Lack of consent to participate in the trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-02-18 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
failure rate of molar tubes | 9 months
  measuring failure rate of molar tubes bonded with modified bonding technique

CONTACTS AND LOCATIONS:
Overall Officials: nawar m hasan, BDS, Principal Investigator — MSc student
Locations (1):
- Almina Dental Clinic, Karbala, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vale E Nascimento AE, Bramante FS, Pinzan-Vercelino CR, Pinzan A, Gurgel JA. Resin reinforcement: an alternative approach for direct bonding of molar tubes. J Clin Orthod. 2014 Jul;48(7):436-40. No abstract available. PMID 25127384
- [Background] Pinzan-Vercelino CR, Pinzan A, Gurgel Jde A, Bramante FS, Pinzan LM. In vitro evaluation of an alternative method to bond molar tubes. J Appl Oral Sci. 2011 Jan-Feb;19(1):41-6. doi: 10.1590/s1678-77572011000100009. PMID 21437468
- [Derived] Hasan NM, Yassir YA. Evaluation of failure rate of molar tubes with a modified bonding technique: a randomized clinical trial. Eur J Orthod. 2023 Nov 30;45(6):764-772. doi: 10.1093/ejo/cjad029. PMID 37467348